CLINICAL TRIAL: NCT06794658
Title: DETERMINATION OF THE EFFICACY OF REMOTE MONITORING OF PATIENTS WITH DIABETES UNDER INSULIN TREATMENT, BY USING Caaring(r) SOFTWARE
Brief Title: EFFICACY OF REMOTE MONITORING OF PATIENTS WITH DIABETES UNDER INSULIN TREATMENT, BY USING Caaring SOFTWARE
Acronym: GluCaaring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Persei Vivarium (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GluCaaring
Record Dates: First submitted 2024-12-17; First posted 2025-01-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus (DM); Remote patient monitoring; glycemic control; Caaring; Time in Range (TIR); Online telemonitoring; Digital Health; DTx; PROMs; Patient-reported data; real-world data
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online telemonitoring group (G_CAARING) (Active Comparator): The monitoring and control of these patients will be carried out remotely through the Caaring® platform. Patients will connect to an APP on a mobile phone. They will have to complete the data and questionnaires related to the study variables.
  Interventions: Device: software
- Retrospective Control group (No Intervention): The data of these patients are collected retrospectively from the medical history, from the last 12 weeks prior to their inclusion.

INTERVENTIONS:
Device: software — Caaring is an electronic data collection notebook that allows patients to confidentially fill out data/questionnaires on their mobile phone and report them through an application that will be installed on the patient's mobile phone. Besides, This group (G_CAARING) will receive educational and prevention recommendations relative to diabetes.
  Other Names: Caaring
  Arms: Online telemonitoring group (G_CAARING)

SUMMARY:
The goal of this clinical trial investigation with device is to determinate the efficacy of the remote monitoring in insulin-treated diabetic patients with a software called Caaring®.

The main question it aims to answer is if the development of a self-management platform (Caaring®) that enhances the role of the patient with diabetes in the course of their disease will increase the TIR and/or reduce the number of in-person and telephone visits assisted by specialized medical and nursing personnel.

This is two arms, randomized study. Online telemonitoring group: The follow-up of these patients will be carried out prospectively remotely through the Caaring® platform. And Retrospective Control group: The data of these patients are collected retrospectively from the last 12 weeks prior to their inclusion.

Researchers will compare the assessments between the two groups to see if the software Caaring® improve the TIR and/or reduce the number of visits to the specialist personnel.

Participants with diabetes will:

Use of continuous subcutaneous insulin infusion (CSII) and continuous glucose monitoring (CGM) systems. In addition,

Control group patients must have clinical and glucometry data from the 12 weeks prior to their inclusion date available in the Medical Record, and/or through the monitoring platforms of the continuous glucose monitoring devices Caaring group patients must have sufficient technological skills to use a smartphone.

DETAILED DESCRIPTION:
This is a longitudinal, comparative non-inferiority, multicenter, with 2 arms Medical Device Clinical Trial.

The protocol and informed consent documents have been reviewed and approved by the hospital human subjects reviewboard and the study will be performed in accordance with the Declaration of Helsinki

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus treated with insulin.
* Patients treated with subcutaneous insulin in multiple daily doses or patients treated with subcutaneous insulin in continuous subcutaneous infusion systems
* Patients using a glucose monitoring system
* Patients who are able to complete the study questionnaires
* Informed consent is obtained from the patient.
* For Control group: Patients must have clinical and glucometry data from the 12 weeks prior to their inclusion date available in the Medical Record, and/or through the monitoring platforms of the continuous glucose monitoring devices - For Caaring group: Patients must have sufficient technological skills to use a smartphone.

Exclusion Criteria:

* Patients with cognitive or sensory difficulties or with insufficient command of Spanish who, in the opinion of the investigator, makes it difficult to understand the questions or the scales, as long as they do not have a legally authorized representative capable of participating in the study.
* Transient patients in whom it may be anticipated that follow-up will not be completed due to a change of residence.
* Patients Who are participating at the time of recruitment in any other clinical trial. Participation in observational studies will not be an exclusion criteria.
* Patients whose main diagnosis is a poorly controlled mental disorders or other medical illness.
* Patients with terminal illness and/or in palliative care according to the criteria of the SECPAL (Spanish Society of Palliative Care).
* Institutionalized patients
* Patients who are pregnant or breastfeeding.
* Patients whose inclusion is not considered advisable by the investigator's assessment due to they are under specific follow-up in other hospital units (hemodialysis, transplants, etc.) that require mandatory hospital attendance less frequently than once every two months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Determinate the efficacy of the remote monitoring in insulin-treated diabetic patients with a software called Caaring®. | 12 weeks
  % acceptable Time in Range (TIR) of glucose measurements defined as the percentage of how long the patient's glucose value was within the target range (70-180 mg/dL)

SECONDARY OUTCOMES:
PROs. Changes in Health-related quality of life (HRQOL): EsDQOL | Day 0 and week 12
  Change in the patient's quality of life scale the study compared to baseline: EsDQOL questionnaire for adults (Value 0-100). A higher score reflects a higher health-related quality of life (HRQoL).
PROs. in Health-related quality of life (HRQOL): KINDL | Day 0 and week 12
  Change in the patient's quality of life scale the study compared to baseline: KINDL and Diabetes-related quality of life questionnaire for pediatrics for the pediatric population (Value 0-100). A higher score reflects a higher health-related quality of life (HRQoL).
PROs. Patient satisfaction with the software Caaring | Week 12
  The patient satisfaction will be measured through a specific satisfaction questionnaire created for this purpose. (Value 3-15). A higher score reflects greater satisfaction with software care.
PROs. Variation in clinical parameters of glycemic control: HbA1c | Day 0 and Week 12
  Variation in clinical parameters of glycemic control, HbA1c
PROs. Variation in clinical parameters of glycemic control, HbA1c and CGM data: TIR | Day 0 and Biweekly up to 12 weeks
  Variation in clinical parameters of glycemic control, HbA1c and CGM data: TIR (time in range)(70-180 mg/dl)
PROs. Variation in clinical parameters of glycemic control, HbA1c and CGM data: TBR | Day 0 and Biweekly up to 12 weeks
  Variation in clinical parameters of glycemic control, HbA1c and CGM data: TBR (time below range) Time < 70 mg/dL
PROs. Variation in clinical parameters of glycemic control, HbA1c and CGM data: TIT | Day 0 and Biweekly up to 12 weeks
  Variation in clinical parameters of glycemic control, HbA1c and CGM data: TIT (Time in target range), (70-140 mg/dL).
PROs. Variation in clinical parameters of glycemic control, HbA1c and CGM data: CV | Day 0 and Biweekly up to 12 weeks
  Variation in clinical parameters of glycemic control, HbA1c and CGM data: CV (Coefficient of Variation)
PROs. Variation in clinical parameters of glycemic control, HbA1c and CGM data: GRI | Day 0 and Biweekly up to 12 weeks
  Variation in clinical parameters of glycemic control, HbA1c and CGM data: GRI (Glycemic Risk Index).
PROs. Number of Medical Visits | Day 0 and Monthly up to 12 weeks
  Number of medical visits, calls or interactions with specialist healthcare personnel
PROs. Adherence of treatment | Day 0 and Weekly up to 12 weeks
  Adherence to therapy (insulin)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Clínico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No